CLINICAL TRIAL: NCT02830633
Title: Trial to Evaluate Laparoscopy-assisted Nerve-preserved Total Mesorectal Excision (LNTME) Versus Open TME for Rectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Han-Hui YAO, M.D., Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LNTME-01
Record Dates: First submitted 2016-06-12; First posted 2016-07-13 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Rectal Cancer
Keywords: laparoscopy; rectal cancer; pelvic autonomic nerve
MeSH Terms: conditions — Rectal Neoplasms

ARMS (2):
- LNTME (Experimental): Laparoscopy-assisted nerve-preserved TME (LNTME) is conducted in rectal cancer patients
  Interventions: Procedure: LNTME
- OTME (Active Comparator): Open TME (OTME) is conducted in rectal cancer patients
  Interventions: Procedure: OTME

INTERVENTIONS:
Procedure: LNTME — Patients in this group received laparoscopy-assisted nerve-preserved TME for treatment of rectal cancer
  Arms: LNTME
Procedure: OTME — Patients in this group received traditional open TME for treatment of rectal cancer
  Arms: OTME

SUMMARY:
The purpose of this study is to determine: (1) whether laparoscopy-assisted nerve-preserved total mesorectal excision (LNTME) is as safe as open TME for rectal cancer, and (2) whether LNTME is more effective for protection of pelvic autonomic nerve function from surgical impairing when comparing to open TME.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients
2. From 18 years old to 60 years old
3. Normal sexual function
4. Tumor located in rectum (defined as 5- to 12-cm from the anal verge)
5. Pathological confirmed rectal cancer
6. Preoperative T stage ranging from T1 to T4a according to the 7th Edition of AJCC Cancer Staging Manual
7. Tumor size < 5 cm
8. ASA score was I-II
9. Informed consent was written

Exclusion Criteria:

1. Distant cancer metastasis
2. History of abdominal surgery
3. With other type of malignancy
4. Preoperative voiding dysfunction
5. Preoperative sexual dysfunction
6. Refusing to attend this trial

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Postoperative complications including bleeding, anastomotic leakage, postoperative infection, organ dysfunctions. | postoperative 30 days
The postoperative sexual function assessed by IIEF questionnaire | postoperative one year
The postoperative voiding function assessed by IPSS questionnaire. | postoperative one year

SECONDARY OUTCOMES:
Operative time | an expected average of 180 minutes
Postoperative deaths | postoperative 30 days
The length postoperative hospital stay | an expected average 8 days
C-reactive protein | postoperative 7 days
  serum C-reactive protein level after operation

REFERENCES:
- [Derived] He Y, Zhu Z, Liu S, Liu L, Hu B, Wan X, Huang Q. [Effect of anastomotic reinforcing sutures on the incidence of anastomotic leakage after laparoscopic radical resection of rectal cancer: a prospective randomized controlled trial]. Zhonghua Wei Chang Wai Ke Za Zhi. 2018 Apirl 25;21(4):431-436. Chinese. PMID 29682715